CLINICAL TRIAL: NCT05071651
Title: Caractéristiques épidémiologiques et méthodes de prévention Des Ampoules Chez Les Coureurs d'Ultra-trail
Brief Title: Epidemiological Characteristics and Prevention Methods of Blisters in Ultra-trail Runners
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Formation et de Recherche en Médecine de Montagne (Other)
Responsible Party: Sponsor
Other Study IDs: Blisters-stop 1
Record Dates: First submitted 2021-08-23; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-08

CONDITIONS: Sport Injury; Blister of Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PRIMARY OBJECTIVE : To evaluate the methods of prevention of the appearance of blisters set up by the runners before and during an ultra-trail

SECONDARY OBJECTIVES :

To evaluate :

* The main locations of blisters.
* The severity of blisters
* The effectiveness of prevention methods To evaluate the incidence of blisters in an ultra-trail context.

DETAILED DESCRIPTION:
MAIN JUDGEMENT CRITERIA :

Prevention methods used before an ultra-trail via a self-questionnaire

SECONDARY JUDGING CRITERIA : Location of blisters, via a self-questionnaire Presence or not of blisters at the end of the ultra-trail or at the time of abandonment

STUDY SCHEME : Post-race questioning

ELIGIBILITY:
Inclusion Criteria:

* Ultra-trail participants with validated registration

Exclusion Criteria:

* Presence of blisters or other skin lesions on the feet before the race

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ultra runners
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Prevention methods used before an ultra-trail via a self-questionnaire | Through study completion, an average of 1 year
  Prevention methods used before an ultra-trail

SECONDARY OUTCOMES:
Location of blisters, via a self-questionnaire | Through study completion, an average of 1 year
  Location of blisters on the feet
Presence or not of blisters at the end of the ultra-trail or at the time of abandonment | Through study completion, an average of 1 year
  Presence or not of blisters at the end

CONTACTS AND LOCATIONS:
Overall Officials: Corentin Tanné, MD, Principal Investigator — Institut de Formation et de Recherche en Médecine de Montagne
Locations (1):
- Ifremmont, Chamonix, France

IPD SHARING:
Plan to Share IPD: No